CLINICAL TRIAL: NCT06413849
Title: Telephone-coached "Graphic Narrative" Bibliotherapy for Informal Caregivers of People With Dementia
Brief Title: Telephone-coached "Graphic Narrative" Bibliotherapy for Dementia Caregivers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: P0047108
Record Dates: First submitted 2024-05-09; First posted 2024-05-14 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2024-05

CONDITIONS: Dementia Caregiver; Depressive Symptoms; Caregiving Appraisal
MeSH Terms: conditions — Depression | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Graphic narrative bibliotherapy (Experimental): Eight weekly sessions of telephone-coached graphic narrative bibliotherapy
  Interventions: Other: Telephone coached graphic narrative bibliotherapy
- Control group (Sham Comparator): Reading an educational booklet
  Interventions: Other: Control group

INTERVENTIONS:
Other: Telephone coached graphic narrative bibliotherapy — Eight weekly sessions of telephone coached graphic narrative bibliotherapy
  Arms: Graphic narrative bibliotherapy
Other: Control group — Reading educational booklet
  Arms: Control group

SUMMARY:
This study aims to assess the efficacy of telephone-coached graphic narrative bibliotherapy in improving dementia caregiver depressive symptoms compared with the booklet group.

DETAILED DESCRIPTION:
This is a two-arm cluster randomized controlled trial using a repeated-measures design to examine the effects of telephone-coached graphic narrative bibliotherapy on 128 (64 per group) informal caregivers of people with dementia. Participants in the intervention group will receive eight weekly telephone-coached graphic narrative bibliotherapy sessions, plus two face-to-face booster sessions and two follow-up sessions. The control group will receive an education booklet and check-in calls. Caregiver depressive symptoms, stress and anxiety, caregiving appraisal, care-recipient neuropsychiatric symptoms, and quality of life will be measured to test the intervention's effects immediately after completion and at a 6-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* provide unpaid care to a person diagnosed with early to moderate stage dementia;
* provide at least 14 hours of care a week for at least 3 months
* aged 18 years or above
* able to read
* have depressive symptoms
* use a message application

Exclusion Criteria:

* with an unstable physical or mental condition
* with cognitive impairment
* receiving medical, psychological, or psychiatric treatment for depression
* have been included in another interventional study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Changes in depressive symptoms | Pre-intervention, immediately post-intervention, 6 months post-intervention
  Depressive symptoms will be measured with the Chinese version of the Depression Anxiety Stress Scale-21. It is a 4-point Likert scale consisting of 21 items that measure levels ofdepression, anxiety, and stress in participants. The total score ranges from 0-63, with the depression subscale score ranges from 0-21. Higher scores indicategreater severity of mental health problems.

SECONDARY OUTCOMES:
Changes in caregiving appraisal | Pre-intervention, immediately post-intervention, 6 months post-intervention
  Caregiving appraisal will be assessed using the Caregiving Appraisal Scale. It is a 26-item Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). The score ranges from 26 to 130. Higher scores on this scale indicate more positive caregiving appraisal.
Changes in stress and anxiety | Pre-intervention, immediately post-intervention, 6 months post-intervention
  Stress and anxiety will be measured with the stress and anxiety subscales of the Depression, anxiety and stress scale-21 (DASS-21). The total score of the full scale ranges from 0-63, with the anxiety and stress subscale score both range from 0-21.
Changes in patient neuropsychiatric symptoms | Pre-intervention, immediately post-intervention, 6 months post-intervention
  Patient neuropsychiatric symptoms: will be measured with the Neuropsychiatric Inventory (NPI). NPI evaluates 12 common neuropsychiatric disturbances in dementia. The presence of problematic behaviors in each domain is assessed by asking an informant a screening question followed by a series of yes/no questions. The frequency of a symptom is created from 1 (rarely) to 4 (very often), and severity is rated from 1 (mild) to 3 (severe).
Changes in quality of life | Pre-intervention, immediately post-intervention, 6 months post-intervention
  Quality of life will be measured with the Brief Older People's Quality of Life Questionnaire (OPQOL-Brief). It is a 13-item, 5-point Likert scale to measure the quality of life for older adults. The total score ranges from 13 to 65, with higher scores indicating a better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong SAR, Hong Kong

IPD SHARING:
Plan to Share IPD: No